CLINICAL TRIAL: NCT05715879
Title: The Long-term Effects of the Covid-19 Infection on Cardiac Symptoms, Should We Have a Realistic Concern?
Brief Title: Covid-19 Infection and Long-term Cardiovascular Symptoms
Status: Completed | Type: Observational
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Other Study IDs: IR.SUMS.MED.REC.1401.465
Record Dates: First submitted 2023-02-04; First posted 2023-02-08 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Pandemic; Dyspnea; Cardiac; Chest Syndrome; Functional Cardiac Disorder
Keywords: Atherosclerosis; covid-19; dyspnea; chest pain
MeSH Terms: conditions — COVID-19; Dyspnea; Atherosclerosis; Chest Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 365 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diseased: covid infection patients
  Interventions: Diagnostic Test: covid infection; Biological: admission to hispital

INTERVENTIONS:
Diagnostic Test: covid infection — patients with covid infection which was proved with positive test
  Other Names: covid 19 infection
Biological: admission to hispital — patients with sever covid disease, who was admitted in hospital

SUMMARY:
From the registry of professor Kojuri clinic , those with Covid-19 infection were selected and was contacted and asked about the cardiovascular symptoms, 1 year after the covid infection

DETAILED DESCRIPTION:
This retrospective cohort study was conducted between October 2020 to May 2021. The study population was patients referring to Professor Kojuri Cardiovascular Clinic in Shiraz, Iran (email: kojurij@yahoo.com, webpage: http://kojuriclinic.com). A database of patients' information is available, including underlying diseases, signs and symptoms, medications, laboratory tests, electrocardiography, and echocardiography. The data is documented by expert cardiologists on every patient's visit.

The inclusion criteria were having a history of COVID-19 infection confirmed by PCR or suggested by HRCT findings and having been afflicted with COVID-19 at least one year ago. The exclusion criteria were having a history of documented COVID-19 infection, which occurred less than a year ago, and having a probable history of COVID-19 not confirmed by PCR or HRCT.

Patients' information before COVID-19 infection was extracted from the database, including baseline demographic data, COVID-19 vaccination history, hypertension (HTN), dyslipidemia (or hyperlipidemia (HLP)), diabetes mellitus (DM), smoking, CVD, and prescribed medications. Patients with incomplete data before COVID-19 or with outdated data were excluded.

We contacted the enrolled patients to get informed about their symptoms, such as dyspnea at rest, dyspnea on exertion (DOE), orthopnea, paroxysmal nocturnal dyspnea (PND) 21, chest pain (CP) 22, fatigue 23, and palpitations 24. Patients were asked to rate their dyspnea at rest from 0 to 10, according to the 10-category ratio. A score of zero means no breathing discomfort, and ten indicates the most severe dyspnea. A score between 1 to 4 was considered mild, 5 to 6 moderate, and 7 to 10 severe. We also used functional class 1 to 4 to assess their dyspnea. Functional class 1 means no limitations in daily activities, functional class 2 means mild exertional dyspnea, functional class 3 indicates moderate dyspnea with daily activities, and functional class 4 figures dyspnea at rest 25. Chest pain was defined, based on the American heart association 2021, as "noncardiac," "possible cardiac," and "cardiac" 22.

A history of major adverse cardiovascular events (MACE) during a year follow-up of COVID-19 infection and admission due to COVID-19 were also reported. MACE is defined as myocardial infarction (MI), admission due to heart failure (HF), stroke, cardiac death, and revascularization procedures, including coronary artery bypass graft (CABG) and percutaneous coronary intervention (PCI) 26.

HTN is defined as clinic SBP ≥140 mm Hg or DBP ≥90 mm Hg in repeated assessment 27. DM is diagnosed based on the American diabetes association (ADA) 2020 guidelines 28. Dyslipidemia is defined as abnormalities in TG, LDL, or HDL cholesterol. A TG level of more than 150 mg/dL is considered abnormal. HDL less than 40 mg/dL, LDL more than 100mg/dL, or is defined as dyslipidemia 29. Current smokers are defined as those who have smoked ≥100 cigarettes and smoked during the 30 days preceding the study. Former smokers have stopped smoking more than 30 days before the research 30.

Statistical analysis was performed using SPSS for Windows ver. 26 (IBM Corp., Armonk, NY, USA). We described continuous variables by mean ±standard deviation. Categorical variables were described by frequency and percentage. We used repeated measure ANOVA and paired-sample t-test for normal distribution variables and Wilcoxon signed-rank test for repeated categorical variables. Pearson's chi-squared test and Kruskal-Wallis test are applied to categorical data. We controlled the effects of confounding factors by using generalized linear models and repeating analyses by different subgroups. Statistical significance was indicated when P<0.05.

All patients were informed about the details of this research and provided their informed consent. Patients who declined to participate in the study were excluded

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infection confirmed by PCR or suggested by HRCT findings and having been afflicted with COVID-19 at least one year ago

Exclusion Criteria:

* COVID-19 infection, which occurred less than a year ago,
* probable history of COVID-19 not confirmed by PCR or HRCT

Ages: 15 Years to 78 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population was patients referring to Professor Kojuri Cardiovascular Clinic in Shiraz, Iran (email: kojurij@yahoo.com, webpage: http://kojuriclinic.com). A database of patients' information is available, including underlying diseases, signs and symptoms, medications, laboratory tests, electrocardiography, and echocardiography. The data is documented by expert cardiologists on every patient's visit.
Sampling Method: Non-Probability Sample
Enrollment: 879 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
dyspnea | 1 year
  Abnormal shortness of breath with lower activities or at rest
chest pain | 1 year
  cheat pain mimicking angina
MACE | 1 year
  major adverse cardiac events, myocardial infarction, admission, death or nead for revascularization

SECONDARY OUTCOMES:
fatigue | 1 year
  feeling weakness with less than ordinary activities

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Ward Shiraz University of Medical Sciences, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Golchin Vafa R, Heydarzadeh R, Rahmani M, Tavan A, Khoshnoud Mansorkhani S, Zamiri B, Amiri F, Azadian A, Khademolhosseini A, Montaseri M, Hosseini N, Hosseini SA, Kojuri J. The long-term effects of the Covid-19 infection on cardiac symptoms. BMC Cardiovasc Disord. 2023 Jun 6;23(1):286. doi: 10.1186/s12872-023-03322-8. PMID 37280530